CLINICAL TRIAL: NCT05335824
Title: Comparison Between The Effect of Platelet Rich Plasma (PRP) and Injectable Platelet Rich Fibrin (I-PRF) on Orthodontic Tooth Movement
Brief Title: The Effect of Autologous Platelet Concentrations on Orthodontic Treatment Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHDS-Ortho-07-2022
Record Dates: First submitted 2022-04-08; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Platelet-rich plasma; Platelet-rich fibrin; Acceleration
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — proliferation regulatory factors, human urine; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The platelet-rich plasma (PRP) group: (Experimental): The patients in this group received PRP injections immediately before the canine retraction, and after 8 weeks of the onset of retraction
  Interventions: Other: The platelet-rich plasma (PRP)
- The injectable platelet-rich fibrin (I-PRF) group (Experimental): The patients in this group received I-PRF injections immediately before the canine retraction, and after 8 weeks of the onset of retraction
  Interventions: Other: The injectable platelet-rich fibrin (I-PRF) group
- The control group (Active Comparator): The patients in this group did not receive any injections
  Interventions: Device: The control group

INTERVENTIONS:
Other: The platelet-rich plasma (PRP) — Twenty ml of venous blood was drawn from each patient with the use of PRP tubes that contain anticoagulant citrate dextrose. The double-spin technique was used to prepare the PRP. The injection areas were anesthetized with lidocaine 2% with epinephrine 1/80000 and left for 10 minutes. 15 units (0. 15 mL) of PRP were injected interaligamentlly in the middle, distobuccal, and distopalatal areas of the distal surface of the upper canines (5 units in each area) together with submucosal injections buccally and palatally (100 units and 50 units
  , respectively).
  Arms: The platelet-rich plasma (PRP) group:
Other: The injectable platelet-rich fibrin (I-PRF) group — Twenty ml of venous blood was drawn from each patient in this experimental group.
  I-PRF was prepared with the use of 20 ml of blood drawn from the patient in dry sterile tubes without anticoagulant (quickly before coagulation starts) by following the centrifugation protocol requires one cycle only (700 RPM for 3 minutes) Injection procedures, sites, and time were similar to the PRP group.
  Arms: The injectable platelet-rich fibrin (I-PRF) group
Device: The control group — NiTi closed-coil springs (American Orthodontics, Sheboygan, WI) were used to impose 150 g force from the first molar band hook to the bracket of canine on each side on 0.019*0.025-in SS archwire Patients' follow-up appointments were two weeks intervals; at each visit, the force produced by the coil was checked and readjusted when needed in order to keep it at 150-g level and the appliances were examined for any deformation or change in the position because of chewing. Canine retraction continued until achieving Class I canine relationship.
  Arms: The control group

SUMMARY:
60 patients needed therapeutic extraction of the maxillary first premolars with subsequent retraction of the maxillary canines were divided to randomly three groups:

(1) PRP group: Received PRP injections, (2) I-PRF group: Received I-PRF injections, (3) Control group: conventional treatment with no injections. TPAs were used as an anchor unit. Coil springs were used to distalize the upper canines on 0.019 x 0.025-inch stainless archwires. Alginate impressions and dental casts of the maxillary arch were done at five-time points over a 4-month follow-up period. The amount of canine movement, canine rotation, and anchorage loss were measured on three-dimensional digital models superimposed on the rugae area.

DETAILED DESCRIPTION:
One of the most important goals of orthodontic treatment is to decrease the treatment time via achieving faster tooth movement chiefly in adults. Adults have more bone density and less bone turnover than adolescence, which may be linked to potential root resorption, periodontal problems, and white spot lesions.

Approaches to reduce orthodontic treatment time included surgical and non-surgical techniques. Non-surgical approaches such as systemic and local administration of chemical substances, low-level laser therapy, vibrations, and pulsed electrical stimulation therapy still need more studies to determine their safety and effectiveness.

Surgical procedures such as corticotomy, corticision, and micro-osteoperforations have

, in general high success rates, but they rely on incurring an injury to bone tissues. The latter has been linked to the regional acceleratory phenomenon (RAP). But the invasive nature of these procedures, associated risks of loss of alveolar bone and gingival recession, and the help needed from another specialist limit its routine application. Recently, the possibility of using platelet-based preparations from the patient's blood to accelerate orthodontic tooth movement like platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) has grown. PRF represents the second generation of biological materials derived from blood. It is obtained through a centrifuge of the patient's blood without adding any additives to the tube. The variety of growth factors in PRP and PRF may have the ability to stimulate the activation of osteoblasts and osteoclasts together, which supports the idea that PRP could affect orthodontic tooth movement The study sample consisted of 60 patients and was calculated using (G-power sample size calculator), depending on the rate of canine retraction with a study power of 90%.

After ensuring the patient's compliance with the terms and conditions of this study, the purpose and methods of the study were explained to the patients using Information Sheet. In case of approval to participate, the patients were asked to sign the informed consent. Extra & Intra-oral photographs, impressions and clinical examinations were made.

Canine retraction was initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. both male and female subjects
2. 18-25 years old
3. Class II Division 1 malocclusion, treated with extraction of the maxillary first premolars
4. Full permanent dentition
5. Good general and oral health

Exclusion Criteria:

1. extreme skeletal class II malocclusion, overjet > 10 mm ANB>7◦
2. diseases and medications that were likely to affect bone biology
3. poor oral hygiene
4. previous orthodontic treatment
5. smoking
6. coagulation disorders, or being treated with anticoagulants

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Change in canine retraction rate | The estimation took place at five time points: the beginning of tooth movement (T0) and at 4, 8, 12, and 16 weeks following T0
  The amount of canine retraction per month was calculated by measuring the distance from the canine cusp tip in the baseline model to the canine cusp tip in the next superimposed model. The amount of distance being retracted in millimeters was divided to the duration of retraction in months to give an estimation of the retraction rate.

SECONDARY OUTCOMES:
Change in the maxillary first molar position (anchorage loss) | T0: before the beginning of canine retraction; T1: after 4 weeks of retraction; T2: after 8 weeks of retraction; T3: after 12 weeks; and T4: after 16 weeks after the start of retraction
  Anchorage loss was calculated in the superimposed digital models from the mesial central fossa of a maxillary first molar of the baseline model the mesial central fossa of maxillary first molar in the next superimposed model.
Change in canine rotation | T0: before the beginning of canine retraction; T1: after 4 weeks of retraction; T2: after 8 weeks of retraction; T3: after 12 weeks; and T4: after 16 weeks after the start of retraction
  The amount of canine rotation was measured in superimposed digital models. Mesial and distal contact points of the canines were used to make a horizontal line that would make an angle with the similar line in the next superimposed model, this angle referred to the amount of canine rotation between the two superimposed models.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ammar, DDS, MSc, Principal Investigator — Department of orthodontics, Hama University, Syria; Rabab al-Sabbagh, DDS,MSc,PhD, Study Director — Department of orthodontics, Hama University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rashid A, ElSharaby FA, Nassef EM, Mehanni S, Mostafa YA. Effect of platelet-rich plasma on orthodontic tooth movement in dogs. Orthod Craniofac Res. 2017 May;20(2):102-110. doi: 10.1111/ocr.12146. PMID 28414871
- [Background] Tehranchi A, Behnia H, Pourdanesh F, Behnia P, Pinto N, Younessian F. The effect of autologous leukocyte platelet rich fibrin on the rate of orthodontic tooth movement: A prospective randomized clinical trial. Eur J Dent. 2018 Jul-Sep;12(3):350-357. doi: 10.4103/ejd.ejd_424_17. PMID 30147398
- [Background] Reyes Pacheco AA, Collins JR, Contreras N, Lantigua A, Pithon MM, Tanaka OM. Distalization rate of maxillary canines in an alveolus filled with leukocyte-platelet-rich fibrin in adults: A randomized controlled clinical split-mouth trial. Am J Orthod Dentofacial Orthop. 2020 Aug;158(2):182-191. doi: 10.1016/j.ajodo.2020.03.020. Epub 2020 Jun 24. PMID 32591274
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Background] Ali Mahmood TM, Chawshli OF. The Effect of Submucosal Injection of Plasma-Rich Platelets on Blood Inflammatory Markers for Patients with Bimaxillary Protrusion Undergoing Orthodontic Treatment. Int J Inflam. 2019 Oct 1;2019:6715871. doi: 10.1155/2019/6715871. eCollection 2019. PMID 31662844
- [Background] Dixon V, Read MJ, O'Brien KD, Worthington HV, Mandall NA. A randomized clinical trial to compare three methods of orthodontic space closure. J Orthod. 2002 Mar;29(1):31-6. doi: 10.1093/ortho/29.1.31. PMID 11907307
- [Derived] Ammar AM, Al-Sabbagh R, Hajeer MY. Evaluation of the effectiveness of the platelet-rich plasma compared to the injectable platelet-rich fibrin on the rate of maxillary canine retraction: a three-arm randomized controlled trial. Eur J Orthod. 2024 Jan 1;46(1):cjad056. doi: 10.1093/ejo/cjad056. PMID 37796117